CLINICAL TRIAL: NCT04688476
Title: An Extended Follow-Up Study of the HPV Vaccine Delayed Booster Trial
Status: Active, not recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sherry Chow, Principal Investigator, University of Arizona
Other Study IDs: 2007882387; UG1 242596 (Other Grant/Funding Number: DCP)
Record Dates: First submitted 2020-12-17; First posted 2020-12-30 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: HPV-associated Cancer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum will be collected at each visit for Serologic geometric mean titers (GMT) of the nine vaccine types (HPV 16/18/ 6/11/31/33/45/52/58).
  Urine will be collected at each visit to explore the potential of assessing HPV DNA and antibodies in the urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is an extended follow-up study to follow-up study participants who received 1 booster dose of Gardasil 9 in the "HPV vaccine delayed booster trial." This was a prospective, single-arm, open-label, non-randomized, phase IIa trial among 9-11 year-old girls and boys to determine the immunogenicity after a single dose of the nonavalent HPV vaccine (Gardasil 9) over 24 months, with a delayed booster dose at 24 months and an optional booster at 30 months after the first dose. Participants provided blood specimens at 6, 12, 18, 24, and 30 months after the first dose. Serologic geometric mean titers (GMT) of the nine vaccine types (HPV 16/18/ 6/11/31/33/45/52/58) were measured at each time point. One hundred and thirty-three (133) participants received one booster dose at month 24 and elected not to receive the second booster at month 30.

For this follow-up study, we anticipate that we will be able to accrue 120 participants from the original study who received just one booster dose. Participants who received one booster dose of Gardasil 9 will be contacted to return to the clinic to provide blood specimens at 48 (±3), 60 (±3), and 72 (±3) months after the priming dose. Serologic geometric mean titers (GMT) of the nine vaccine types (HPV 16/18/ 6/11/31/33/45/52/58) will be measured at each time point.

ELIGIBILITY:
Inclusion Criteria:

* Study participants who received one booster dose of Gardasil 9 at month 24 and elected not to receive the second booster at month 30 in the original "HPV vaccine delayed booster trial"
* Ability to understand and the willingness to sign a written informed consent document by the legal representative(s) of the participant.
* Ability to understand and the willingness to sign a written assent document by the participant.

Exclusion Criteria:

- Has received any HPV vaccine dose from an external source at any point during or after participation in the HPV vaccine delayed booster trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Study population is restricted to study participants who received one booster dose of Gardasil 9 at month 24 and elected not to receive the second booster at month 30 in the original "HPV vaccine delayed booster trial".
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The differences in geometric mean titer (GMT) of HPV 16 and HPV18 between 30 vs. 48, 48 vs. 60, and 60 vs. 72 months after the priming dose of Gardasil | 72 months

SECONDARY OUTCOMES:
The differences in geometric mean titer of other HPV types (HPV6/11/31/33/45/52/58) between 30 vs. 48, 48 vs. 60, and 60 vs. 72 months after the priming dose of Gardasil 9 | 72 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Arizona, Tucson, Arizona
  - University of California, Los Angeles, Los Angeles, California

IPD SHARING:
Plan to Share IPD: No